CLINICAL TRIAL: NCT05517265
Title: A Non-interventional, Prospective, Open-label, Observational Study Evaluating the Effectiveness and Safety of Acalabrutinib (Calquence®) in Patients With Chronic Lymphocytic Leukemia (CLL) Receiving Direct Oral Anticoagulation (DOAC).
Brief Title: Acalabrutinib in Patients With Chronic Lymphocytic Leukemia With Direct Oral Anticoagulation (CICERO)
Acronym: CICERO
Status: Active, not recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-100473
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: CLL
Keywords: CLL; Acalabrutinib (+/- Obinutuzumab); DOAC
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- first-line therapy: Patients enrolled for first-line acalabrutinib (+/- obinutuzumab).
  Interventions: Drug: Calquence
- later-line therapy: Pre-treated patients enrolled for later-line acalabrutinib therapy.
  Interventions: Drug: Calquence

INTERVENTIONS:
Drug: Calquence — acalabrutinib (+/- obinutuzumab) according to Calquence® SmPC.
  Groups: first-line therapy
Drug: Calquence — acalabrutinib according to Calquence® SmPC.
  Groups: later-line therapy

SUMMARY:
The goal of CICERO is to investigate the clinical outcome with a particular focus on prospective data on safety using acalabrutinib (+/- obinutuzumab) in CLL patients receiving co-medication with DOACs (edoxaban, rivaroxaban, dabigatran, apixaban) irrespective of treatment line.

DETAILED DESCRIPTION:
The non-interventional study (NIS) CICERO will collect real-world data to explore acalabrutinib (+/- obinutuzumab) in adult CLL patients (irrespective of treatment line) who receive co-medication with DOACs. The primary focus of the study is to investigate the incidence proportion of bleeding events. Due to the mostly elderly CLL patient population, CLL patients often suffer from multiple cardiovascular comorbidities including atrial fibrillation (AF), deep vein thrombosis (DVT) or pulmonary embolism (PE) which make anticoagulation mandatory.

Up to now, no systematic and prospective evaluation on interactions of BTKis and DOACs has been conducted.

In Order to assess bleeding events, a questionnaire will be used to document if bleeding events occurred in-between visits in routine care. Patients will be asked at each visit if distinct events occurred in the time between the last visit until the current visit and discuss the questionnaire with the physician to determine of any (S)AE occurred until end of acalabrutinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with chronic lymphocytic leukemia (CLL) and decision for treatment with acalabrutinib (+/- obinutuzumab) according to current SmPC as assessed by the treating physician or already started treatment with acalabrutinib (+/- obinutuzumab) according to current SmPC no longer than 6 weeks ago
* Other concomitant disease resulting in medical need of or already under treatment with direct oral anticoagulant (DOAC) treatment with edoxaban (Lixiana®) or rivaroxaban (Xarelto®) or dabigatran (Pradaxa®) or apixaban (Eliquis®) according to the respective current SmPC.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Signed, written informed consent.

Exclusion Criteria:

* Combination of acalabrutinib with other substances than obinutuzumab for CLL treatment
* Participation in an interventional clinical trial with acalabrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with CLL receiving acalabrutinib (+/- obinutuzumab) and co-medication with DOAC.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence proportion of patients with major bleeding event according to Schulman et al. | Baseline until end of acalabrutinib treatment (+ 30 days safety follow-up); up to 41 months
  Bleeding event is defined as major according to Schulmann et al., if it is fatal (contributes to death) and/or symptomatic in a critical area or organ (such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome) and/or causing a decrease in hemoglobin of 2 g/dL (1.24 mmol/l) or more or requires a transfusion of 2 or more units of whole blood or red blood cells.
  Incidence proportion (cumulative incidence) is calculated as the number of patients with bleeding event while on treatment (+30 days safety follow-up), divided by the number of patients in the full analysis population.

SECONDARY OUTCOMES:
Incidence proportion of clinically relevant non-major (CRNM) bleeding events | Baseline, up to 41 months
  CRNM bleeding is defined as bleeding that does not meet the criteria for major bleeding according to Schulman et al. but is associated with the need for medical intervention and/or personal contact with a physician and/or hospitalization or increase in level of care.
Major (according to Schulman et al.) and/or CRNM bleeding events. | Baseline, up to 41 months
  Incidence proportion of major (according to Schulman et al.) and/or CRNM bleeding events.
Any bleeding event. | Baseline, up to 41 months
  Incidence proportion of any bleeding event.
Incidence proportion of major bleeding according to Ghia et al. | Baseline, up to 41 months
  Major bleeding according to Ghia et al. is defined as any serious OR grade ≥3 hemorrhage OR central nervous system (CNS) hemorrhage of any grade, excluding immune thrombocytopenic purpura.
Time to first Occurrence of major bleeding events | Baseline, up to 41 months
  Time to first occurrence of major (according to Schulman et al.) bleeding events.
Incidence proportion of central nervous system (CNS) bleeding events | Baseline, up to 41 months
  Frequencies of patients with CNS bleeding events.
Patient safety regarding mortality | Baseline, up to 41 months
  Mortality from all causes during acalabrutinib therapy.
Patient safety in terms of interactions with effectiveness of DOAC | Baseline, up to 41 months
  Rate of any new or recurrent ischemic stroke or arterial systemic embolism or venous thromboembolic events.
VTE (venous thromboembolism)-related death | Baseline, up to 41 months
  Incidence proportion of VTE-related death.
Overall response rate (ORR) | Baseline, up to 41 months
  ORR is defined as proportion of patients with any response (partial or complete remission) overall.
Progression-free survival (PFS) | Baseline, up to 41 months
  Time from start of acalabrutinib to occurrence of progressive disease or death from any cause, whichever comes first.
Overall survival (OS) | Baseline, up to 41 months
  OS is defined as time from first administration of acalabrutinib to death from any cause.
Therapy decision making | Baseline
  Frequencies of parameters affecting therapy choice.
Previous therapies | Baseline
  Frequencies and percentages of previous therapies
Acalabrutinib (+/- obinutuzumab) treatment: Duration | Baseline, up to 41 months
  Analysis of treatment duration of acalabrutinib using descriptive statistics.
Acalabrutinib (+/- obinutuzumab) treatment: Dose intensity | Baseline, up to 41 months
  Analysis of dose intensity of acalabrutinib treatment with reference to the SmPC (absolute and relative) using descriptive statistics.
Obinutuzumab treatment: Duration | Baseline, up to 41 months
  Analysis of treatment duration of obinutuzumab using descriptive statistics
Reasons for end of treatment of obinutuzumab | Baseline, up to 41 months
  Frequencies and percentages of reasons for end of obinutuzumab treatment.
Types of DOAC | Baseline, up to 41 months
  Type of DOAC used (edoxaban, rivaroxaban, dabigatran and apixaban).
Reasons for DOAC treatment | Baseline, up to 41 months
  Frequencies and precentages of reasons for DOAC treatment.
DOAC treatment: Duration | Baseline, up to 41 months
  Analysis of DOAC treatment duration using descriptive statistics.
DOAC treatment: Dose modifications | Baseline, up to 41 months
  Frequencies and percentages of dose modifications of DOAC treatment.
DOAC treatment: Reasons for dose modifications | Baseline, up to 41 months
  Frequencies and percentages of reasons for dose modifications of DOAC treatment.
DOAC treatment: Reasons for end of treatment | Baseline, up to 41 months
  Frequencies and percentages of reasons for end of DOAC treatment.
Time from onset to DOAC to start of acalabrutinib | Baseline, up to 41 months
  Assessment of time from onset of DOAC to start of acalabrutinib therapy using descriptive statistics.
Concomitant medication | Baseline, up to 41 months
  Frequency of concomitant medication other than DOAC.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Fenchel, Prof. Dr., Study Chair — Onkologische Praxisklinik Hämatologie/ Onkologie und Gerinnungsstörungen
Locations (1):
- Prof. Dr. Fenchel & Dr. Winkler MVZ Träger GbR, Saalfeld, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Ghia P, Pluta A, Wach M, Lysak D, Kozak T, Simkovic M, Kaplan P, Kraychok I, Illes A, de la Serna J, Dolan S, Campbell P, Musuraca G, Jacob A, Avery E, Lee JH, Liang W, Patel P, Quah C, Jurczak W. ASCEND: Phase III, Randomized Trial of Acalabrutinib Versus Idelalisib Plus Rituximab or Bendamustine Plus Rituximab in Relapsed or Refractory Chronic Lymphocytic Leukemia. J Clin Oncol. 2020 Sep 1;38(25):2849-2861. doi: 10.1200/JCO.19.03355. Epub 2020 May 27. PMID 32459600